CLINICAL TRIAL: NCT01759758
Title: Conventional Plaster Versus Thermoplastic Splint for the Treatment of a Pediatric Metacarpal Neck Fracture: a Randomized Trial
Brief Title: A Randomized Trial Comparing Conventional Plaster and Thermoplastic Splints to Treat Pediatric Boxer's Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Michael Bezuhly, Assistant Professor, Clinical Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IWK-1012457
Record Dates: First submitted 2012-12-30; First posted 2013-01-03 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Bone Fractures; Splints; Metacarpal Fracture; Boxer's Fracture
Keywords: boxer's fracture; metacarpal neck fracture; metacarpal fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Calcium Sulfate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plaster Ulnar Gutter Splint (Active Comparator): Patients will have their hand placed in a conventional Plaster ulnar gutter splint. This immobilizes all joints of the ring and small fingers and the wrist
  Interventions: Other: Plaster Ulnar Gutter Splint
- Thermoplastic Splint (Experimental): Patients will be fitted with a custom molded thermoplastic splint that stabilizes the metacarpals of the injured hand but does not immobilize any joints
  Interventions: Other: Thermoplastic Splint

INTERVENTIONS:
Other: Plaster Ulnar Gutter Splint — Patients are placed in a plaster ulnar gutter splint, molded in the safe position.
  Other Names: Conventional Plaster splint; Plaster of Paris
  Arms: Plaster Ulnar Gutter Splint
Other: Thermoplastic Splint — Thermoplastic Splint is heat moulded to the patient's hand, stabilizing the metacarpal heads, but not immobilizing any joints. This is done by our occupational therapist.
  Other Names: Functional brace; Moulded brace; Moulded Metacarpal brace
  Arms: Thermoplastic Splint

SUMMARY:
The investigators are conducting a randomized clinical trial comparing two types of splints for treatment of Boxer's fractures in children up to age 17 inclusive. Patients who meet inclusion criteria will be randomized to either Group A or B. Group A will be treated with the conventional plaster ulnar gutter splint. Group B will be treated with a custom molded thermoplastic hand-based splint. The thermoplastic splint will provide support of the metacarpal but does not immobilize the patient's wrist or interphalangeal joints.

Hypothesis: Is plaster splint immobilization an equivalent treatment method to a custom made thermoplastic splint for a fifth metacarpal neck fracture? Will one splint be tolerated better than the other and will the compliance be different between the two groups?

DETAILED DESCRIPTION:
Nearly all Boxer's fractures are treated without surgery using a splint to keep part or all of the hand from moving (immobilization). There are several acceptable methods of immobilization used by hand surgeons, using splints of different sizes and materials for variable periods of time(1-6).

A recent systematic review from The Cochrane Collaboration found the current data to be inconclusive with regards to the optimal immobilization technique and highlighted the need for further studies(2). Specifically, it was recommended that future studies include functional outcome measures, timing of return to work, complications, pain scores, and an economic analysis.

The current practice at the investigators' institution is for patients to be splinted in a plaster ulnar gutter splint, in the Emergency Department and referred to the next available plastic surgery clinic. If needed, a closed reduction would be performed in clinic, if there was a significant angulation (greater than 45 degrees) or any clinical rotation deformity. The most common method of immobilization involves placing the wrist, ring finger and little finger all the way from the fingertips to the mid-forearm in molded plaster called an ulnar gutter splint. The splint is left on 24 hours a day for 3 to 4 weeks and then removed in the clinic.

Many patients find it difficult to keep the splint on for the full 3 to 4 weeks for a number of reasons. The plaster needs to stay dry, making it awkward to bathe. The splint can also get loose and rub as the swelling around the fracture gets better. The splint can also start to smell because sweat builds up under it. Some patients find the plaster material heavy, making it difficult to wear. Finally, many patients are self-conscious about the appearance of the splint and remove it for this reason alone. In the investigators' experience, up to 1 out of 5 patients will remove the splint on their own against doctor's orders for one reason or another. When patients do follow instructions and keep the splint on 24 hours a day for 3 to 4 weeks, this can lead to joint stiffness when the splint is removed. Some patients may even require physiotherapy to regain their normal finger movement and grip strength.

It is unknown if the ulnar gutter splint is really the best way to immobilize the hand after a Boxer's fracture. It is unknown what material is best for making the splint, whether it is truly necessary to keep the entirety of the wrist and ring and little fingers still, and for how long the hand and fingers should be kept still. Most surgeons recommend patients wear a splint for 3 to 4 weeks.

The investigators would like to determine if a smaller splint made of more durable, lighter moldable plastic that allows earlier movement of the hand and fingers while still keeping the fracture from moving gives the same result as the commonly used ulnar gutter splint.

Functional Hand Based Splint (Thermoplastic Splint) The functional hand-based splint is made of custom molded hard plastic and is fitted over the hand only. A thermoplastic splint is made from plastic that is heated and custom-fitted to the subject's hand, which hardens when it cools. This thermoplastic splint is custom fitted by an occupational therapist such that all joints are free to move. The splint does not limit the patient from moving their wrist or fingers while wearing it. It is custom molded such that it fits snuggly over the patient's hand and holds the fracture in a stable position.

Several adult studies have found this type of custom molded splint superior to either surgical treatment and/or plaster splint immobilization because it resulted in less stiffness, better movement after splint removal, and no increased pain (4-7). The investigators are not aware of any comparative studies done in pediatric patients.

Compliance Patient compliance for wearing their splint for the prescribed during can be a problem. At the investigators' institution, there is a non-compliance rate of approximately 15 to 20 % for Boxer's fracture patients. The investigators hypothesize that the hand-based splint will be better tolerated by patients and therefore result in a higher rate of compliance for the prescribed duration that the plaster splint. Also, the thermoplastic splint will not be damaged if it gets wet, which may translate into fewer additional visits to the clinic or emergency department to have the splint replaced.

This study will be a randomized, single-blinded controlled trial. The randomization of the two splint types will be determined by a computer-based number generator. The patients will know what type of splint they have, but the plastic surgeons and physiotherapist who examine and test the subjects ROM and grip strength will not know the type of splint for each subject.

Patients will be randomized to one of the two groups at their first clinic visit, within 7 days of their injury. They will have their splint placed at this visit and are to wear the splint at all times for 3 weeks. Subjects will return to clinic at 1, 3, 6, and 12 weeks to be reassessed. Specified outcome measures (primary and secondary) will be tested at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Isolated 5th metacarpal neck fracture
* Less than 10 days from injury

Exclusion Criteria:

* Multiple Metacarpal fractures
* Significant injuries to other hand structures (tendons, nerves, major arteries)

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Range of Motion | up to 12 weeks
  The active and passive Range of Motion (ROM) will be tested at 3 time points, for all fingers and the wrist
Compliance | 3 weeks post fracture
  The compliance rate of subjects in each group wearing the splint at all times for the prescribed duration (3 weeks) will be assessed.

SECONDARY OUTCOMES:
Pain | 1, 3, 6, and 12 weeks post fracture
  Pain, reported on a Visual Analog Scale, will be assessed at specified time points
Complications | 3, 6, and 12 weeks
  Loss of fracture reduction, malunion or non-union will be monitored throughout the study
Validated Outcome Questionnaire | 3, 6, and 12 weeks
  Patients will complete the Pediatric Outcomes Data Collection Instrument (PODCI) at several time points
Grip Strength | 6 and 12 weeks
  Patients will have their grip strength measured for the injured and non-injured hand at 6 and 12 weeks post fracture
Radiographic assessment of fracture | 12 weeks post fracture
  An X-ray of the injured had will be done in 3 views. This will be assessed by one of the investigators, in a blinded fashion. They will determine the angulation and assess for evidence of bony healing

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bezuhly, MD, MSc, SM, Principal Investigator — Assistant Professor, Clinician-Investigator at IWK Health Centre and Dalhousie University
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Hunter JM, Cowen NJ. Fifth metacarpal fractures in a compensation clinic population. A report on one hundred and thirty-three cases. J Bone Joint Surg Am. 1970 Sep;52(6):1159-65. No abstract available. PMID 4247878
- [Background] Poolman RW, Goslings JC, Lee JB, Statius Muller M, Steller EP, Struijs PA. Conservative treatment for closed fifth (small finger) metacarpal neck fractures. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD003210. doi: 10.1002/14651858.CD003210.pub3. PMID 16034891
- [Background] Braakman M, Oderwald EE, Haentjens MH. Functional taping of fractures of the 5th metacarpal results in a quicker recovery. Injury. 1998 Jan;29(1):5-9. doi: 10.1016/s0020-1383(97)00106-x. PMID 9659472
- [Background] Harding IJ, Parry D, Barrington RL. The use of a moulded metacarpal brace versus neighbour strapping for fractures of the little finger metacarpal neck. J Hand Surg Br. 2001 Jun;26(3):261-3. doi: 10.1054/jhsb.2000.0509. PMID 11386781
- [Background] Kuokkanen HO, Mulari-Keranen SK, Niskanen RO, Haapala JK, Korkala OL. Treatment of subcapital fractures of the fifth metacarpal bone: a prospective randomised comparison between functional treatment and reposition and splinting. Scand J Plast Reconstr Surg Hand Surg. 1999 Sep;33(3):315-7. doi: 10.1080/02844319950159299. PMID 10505445
- [Background] Statius Muller MG, Poolman RW, van Hoogstraten MJ, Steller EP. Immediate mobilization gives good results in boxer's fractures with volar angulation up to 70 degrees: a prospective randomized trial comparing immediate mobilization with cast immobilization. Arch Orthop Trauma Surg. 2003 Dec;123(10):534-7. doi: 10.1007/s00402-003-0580-2. Epub 2003 Aug 28. PMID 14639483
- [Background] Hansen PB, Hansen TB. The treatment of fractures of the ring and little metacarpal necks. A prospective randomized study of three different types of treatment. J Hand Surg Br. 1998 Apr;23(2):245-7. doi: 10.1016/s0266-7681(98)80186-1. PMID 9607671
- [Background] Konradsen L, Nielsen PT, Albrecht-Beste E. Functional treatment of metacarpal fractures 100 randomized cases with or without fixation. Acta Orthop Scand. 1990 Dec;61(6):531-4. doi: 10.3109/17453679008993576. PMID 2281761
- [Background] Sawyer JR, Ivie CB, Huff AL, Wheeler C, Kelly DM, Beaty JH, Canale ST. Emergency room visits by pediatric fracture patients treated with cast immobilization. J Pediatr Orthop. 2010 Apr-May;30(3):248-52. doi: 10.1097/BPO.0b013e3181d213bc. PMID 20357591
- [Background] Strub B, Schindele S, Sonderegger J, Sproedt J, von Campe A, Gruenert JG. Intramedullary splinting or conservative treatment for displaced fractures of the little finger metacarpal neck? A prospective study. J Hand Surg Eur Vol. 2010 Nov;35(9):725-9. doi: 10.1177/1753193410377845. Epub 2010 Jul 21. PMID 20659966
- [Background] Hofmeister EP, Kim J, Shin AY. Comparison of 2 methods of immobilization of fifth metacarpal neck fractures: a prospective randomized study. J Hand Surg Am. 2008 Oct;33(8):1362-8. doi: 10.1016/j.jhsa.2008.04.010. PMID 18929202
- [Background] Lerman JA, Sullivan E, Barnes DA, Haynes RJ. The Pediatric Outcomes Data Collection Instrument (PODCI) and functional assessment of patients with unilateral upper extremity deficiencies. J Pediatr Orthop. 2005 May-Jun;25(3):405-7. doi: 10.1097/01.bpo.0000149866.80894.70. PMID 15832164
- [Derived] Davison PG, Boudreau N, Burrows R, Wilson KL, Bezuhly M. Forearm-Based Ulnar Gutter versus Hand-Based Thermoplastic Splint for Pediatric Metacarpal Neck Fractures: A Blinded, Randomized Trial. Plast Reconstr Surg. 2016 Mar;137(3):908-916. doi: 10.1097/01.prs.0000479974.45051.78. PMID 26910672